CLINICAL TRIAL: NCT04556955
Title: Comparison of Post Isometric Relaxation and Graston Technique in Mechanical Neck Pain.
Brief Title: The Comparison of PIR and GT in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00683 Sakina Sheikh
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Mechanical Neck Pain
Keywords: Post isometric relaxation; Graston technique; Mechanical neck pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post isometric relaxation and exercises (Placebo Comparator): Group A included Post Isometric Relaxation, 5 rep , 20% isometric contraction 10 sec , 20 sec of stretch hold beyond resistance barrier and conventional exercise program ; this program included Hot pack placed over the painful area in cervical region before the treatment ( 20 minutes).Strengthening exercises for deep neck flexors, rhomboids, lower trapezius and serratus anterior due to weak muscles (2 sets of 10 repetitions once a day) Stretching exercises for pectoralis muscles (20-second hold, 5 repetitions).This exercise protocol was for 4 weeks and 3 sessions per week. Measurements taken at baseline level and at the End of treatment, i.e. ROM, pain intensity by NPRS and PPT , functional disability.
  Interventions: Other: post isometric relaxation
- Graston technique and exercises (Experimental): Group B included Graston Technique to Upper Trapezius and Levator Scapulae.This instrumented-assisted soft tissue massage applied with deeper pressure to the area of concern.The protocol consist of Longitudinal stroking parallel to muscle fiber for 1min , spin over trigger points for 1 min using knob of instrument and fanning for 2 min Hot pack placed over the painful area in cervical region before the treatment ( 20 minutes).Strengthening exercises for deep neck flexors, rhomboids, lower trapezius and serratus anterior due to weak muscles (2 sets of 10 repetitions once a day) Stretching exercises for pectoralis muscles (20-second hold, 5 repetitions). This exercise protocol was for 4 weeks and 3 sessions per week. Measurements taken at baseline level and at the END of treatment , i.e. ROM, pain intensity by NPRS and PPT , functional disability.
  Interventions: Device: Graston technique

INTERVENTIONS:
Device: Graston technique — Experimental group included Graston technique :The protocol consist of Longitudinal stroking parallel to muscle fiber for 1min , spin over trigger points for 1 min using knob of instrument and fanning for 2 min.
  Arms: Graston technique and exercises
Other: post isometric relaxation — Post Isometric Relaxation, 5 rep , 20% isometric contraction 10 sec , 20 sec of stretch hold beyond resistance barrier
  Arms: post isometric relaxation and exercises

SUMMARY:
The aim of this research is to compare the effects of post isometric relaxation and graston technique in mechanical neck pain. Post isometric relaxation and graston effects on pain , cervical range of motion and function. A randomized controlled trial was done at Max health hospital G-8 markaz Islamabad . The sample size was 20. The Participants were divided into two groups,10 participants in group A (post iso metric relaxation) and 10 in group B (Graston technique ) . The study duration was 6 months. Sampling technique applied was purposive sampling technique Randomized through sealed enveloped method . Only 18 to 50 years participants with mechanical neck pain were included in the study . Outcome measure Tools used in this study were Numerical pain rating scale (NPRS) ,inclinometer for cervical ROM, Algometer for pain pressure threshold and Neck disability index for assessing functional disability . Data analyzed through SPSS version 20.

DETAILED DESCRIPTION:
Among all Musculoskeletal disorders occuring in general population ,the neck pain is one of the most common disorder. It's prevalence ranges from 14.2% to 71% in the general population and more prevalent in adult women With the adult age of 15-74 years it's mean point prevalence becomes 7.6%. The child's et al concluded that the life time prevalence of neck pain is 22-70% Among computer workers it has been observed higher incidence , the studies predicted one year incidence of neck pain from 10.4% to 21.3%. Neck pain is defined as "the pain anywhere within the region bounded superiorly by superior nuchal line, inferiorly by an imaginary line through the tip of first thoracic spinous process and laterally by sagittal plane tangential to the lateral borders of the neck"..

Postural and mechanical based symptoms occurs in Mechanical neck pain that are under the influence of many factors that's why difficult to understand.The evidence of studies suggests prolonged adapted posture and repetitive movements falls under the category of biomechanical factors that introduce neck pain whereas according to psychosocial stress associated with neck pain , in which over activity of trapezius muscle motor units monitored , due to increased mental and physical demand of work . That Results in Muscle spasm and pain , majorly caused by long time exposure to these stressors which can lead to functional disability , reduces activity level , anxiety , depression overall influence the quality of life of individual.

Evidence supported by studies that , in subjects with mechanical neck pain may have trigger points in cervical muscles that include upper trapezius , levator scapulae and sternocleidomastoid muscles . When palpated elicited referred pain pattern , so responsible for major provoked symptoms of Mechanical neck pain. In the cervical region the upper trapezius , levator scapulae , scalene and sternocleidomastoid muscles are tend to be more tight and painful thus their lengthening is more prioritized. Along with the upper trapezius is considered as the most commonly involved muscle. The trigger points are defined as the taut bands of skeletal muscle tissues in hypersensitive areas that generates pain on palpation and shows tenderness on touch. In individual with Mechanical neck pain , the pain processes may involve muscular trigger points. According to shah et al it has been shown that Mechanical Neck Pain is associated with sensitization mechanisms, the algogenic substances and chemical mediators (potassium , serotonin, bradykinin ,histamine , prostaglandins and leukotrienes) that involved in tissue damage can also lead to peripheral transduction are present in higher level in active trigger points than latent trigger points.

Literature Review :A Systemic review or Meta-analysis in 2017 by including 7 studies after screening 1169 articles to determine the impact of manual therapy and exercise therapy as combined treatment or delivered alone for the treatment of neck pain patients. They concluded that combined treatment were no more effective for improving outcomes.

In 2018 done a metaanalysis conducted to determine the effects of thoracic manipulation on pain and disability in patients of chronic mechanical neck pain . The results describes that thrust manipulation was highly effective than non thrust manipulation for reducing pain and disability associated with mechanical neck pain patients In 2019 a systemic review of 47 randomized controlled trails studies conducted about treatment of chronic non specific neck pain majorly focused on efficacy , effectiveness and safety of manipulation , mobilization and multi-modal approaches.They also predicted that multi-modal approach may have more impact in decreasing pain and increasing function in patients with non specific neck pain.

The study Results suggested that Adding Post isometric relaxation technique to the conventional physical therapy treatment program of chronic Mechanical Neck Pain was more effective in reducing pain and functional disability and increasing cervical ROM than the traditional treatment program alone.

A study in 2016 suggested that for Muscle energy technique reduces the pain and functional disability higher than stretching technique.

A study suggested that for reducing pain and increasing Range of motion Muscle energy technique was better than static stretching in treating patients with mechanical neck pain.

According to an Randomized controlled trail study that compared the efficacy of spinal manipulative therapy and Graston technique for the treatment of non specific thoracic pain.There is no significant difference in outcome at any point for pain or disability when comparing Spinal manipulative Therapy , Graston Technique.

According to an RCT , the Post Isometric Relaxation was highly beneficial for improving cervical ROM and reducing pain , associated disability in non specific neck pain patients then isometric exercises.

According to comparative study in 2017, results suggested increase in neck mobility and reduction in pain , but concluded that Muscle energy technique was more beneficial than positional release technique in patient's with non-specific neck pain.

In 2016 According to a study in patients with chronic mechanical neck pain .The outcome measure tools was Visual Analogue Scale for pain intensity , universal goniometer used to measure rotation and lateral flexion of neck muscles while function was determined by Neck Disability Index scale. Results showed improvement in both Proprioceptive Neuromuscular facilitation and Muscle Energy Technique .

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of Mechanical neck pain 4-12 weeks.
* Neck pain rating on NPRS (4-8 )
* Palpable pain on Active or latent trigger points

Exclusion Criteria:

* signs of serious pathology (e.g., malignancy, inflammatory disorder, infection)
* history of cervical spine surgery in previous 12 months
* history of trauma or fractures in cervical spine
* signs of cervical radiculopathy
* Vascular syndromes such as basilar insufficiency.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) for pain. | 12th day.
  Numeric Pain Rating Scale (NPRS) for pain : is a unidimensional measure of pain intensity .The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable") Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
Cervical range of motion by using Inclinometer | 12th day
  Measuring Cervical flexion, extension , Right side bending , left side bending , right rotation and Left rotation

SECONDARY OUTCOMES:
Neck disability index for assessing functional status | 12th day
  It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain
Algometry for assessing pressure pain threshold for trigger points. | 12th day
  Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold on trigger points of upper trapezius and levator scapulae.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital., Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Binder AI. Cervical spondylosis and neck pain. BMJ. 2007 Mar 10;334(7592):527-31. doi: 10.1136/bmj.39127.608299.80. No abstract available. PMID 17347239
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Osama M, Shakil Ur Rehman S. Effects of static stretching as compared to autogenic inhibition and reciprocal inhibition muscle energy techniques in the management of mechanical neck pain: a randomized controlled trial. J Pak Med Assoc. 2020 May;70(5):786-790. doi: 10.5455/JPMA.9596. PMID 32400728
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] Misailidou V, Malliou P, Beneka A, Karagiannidis A, Godolias G. Assessment of patients with neck pain: a review of definitions, selection criteria, and measurement tools. J Chiropr Med. 2010 Jun;9(2):49-59. doi: 10.1016/j.jcm.2010.03.002. PMID 21629550
- [Background] Cote P, Cassidy DJ, Carroll LJ, Kristman V. The annual incidence and course of neck pain in the general population: a population-based cohort study. Pain. 2004 Dec;112(3):267-273. doi: 10.1016/j.pain.2004.09.004. PMID 15561381
- [Background] Stephenson JL, Christou EA, Maluf KS. Discharge rate modulation of trapezius motor units differs for voluntary contractions and instructed muscle rest. Exp Brain Res. 2011 Jan;208(2):203-15. doi: 10.1007/s00221-010-2471-4. Epub 2010 Nov 10. PMID 21063691
- [Background] Lundberg U, Kadefors R, Melin B, Palmerud G, Hassmen P, Engstrom M, Dohns IE. Psychophysiological stress and EMG activity of the trapezius muscle. Int J Behav Med. 1994;1(4):354-70. doi: 10.1207/s15327558ijbm0104_5. PMID 16250795
- [Background] Bruflat AK, Balter JE, McGuire D, Fethke NB, Maluf KS. Stress management as an adjunct to physical therapy for chronic neck pain. Phys Ther. 2012 Oct;92(10):1348-59. doi: 10.2522/ptj.20110489. Epub 2012 Jun 14. PMID 22700538
- [Background] Munoz-Munoz S, Munoz-Garcia MT, Alburquerque-Sendin F, Arroyo-Morales M, Fernandez-de-las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in individuals with mechanical neck pain. J Manipulative Physiol Ther. 2012 Oct;35(8):608-13. doi: 10.1016/j.jmpt.2012.09.003. PMID 23158466
- [Background] Mejuto-Vazquez MJ, Salom-Moreno J, Ortega-Santiago R, Truyols-Dominguez S, Fernandez-de-Las-Penas C. Short-term changes in neck pain, widespread pressure pain sensitivity, and cervical range of motion after the application of trigger point dry needling in patients with acute mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Apr;44(4):252-60. doi: 10.2519/jospt.2014.5108. Epub 2014 Feb 25. PMID 24568260
- [Background] Fernandez-de-las-Penas C, Alonso-Blanco C, Miangolarra JC. Myofascial trigger points in subjects presenting with mechanical neck pain: a blinded, controlled study. Man Ther. 2007 Feb;12(1):29-33. doi: 10.1016/j.math.2006.02.002. PMID 21882489
- [Background] Fredin K, Loras H. Manual therapy, exercise therapy or combined treatment in the management of adult neck pain - A systematic review and meta-analysis. Musculoskelet Sci Pract. 2017 Oct;31:62-71. doi: 10.1016/j.msksp.2017.07.005. Epub 2017 Jul 21. PMID 28750310
- [Background] Thornton, C., The effects of thoracic manipulation in the treatment of mechanical neck pain: a meta-analysis. 2018.
- [Background] Coulter ID, Crawford C, Vernon H, Hurwitz EL, Khorsan R, Booth MS, Herman PM. Manipulation and Mobilization for Treating Chronic Nonspecific Neck Pain: A Systematic Review and Meta-Analysis for an Appropriateness Panel. Pain Physician. 2019 Mar;22(2):E55-E70. PMID 30921975
- [Background] • El Laithy, M.H. and K.Z. Fouda, Effect of post isometric relaxation technique in the treatment of mechanical neck pain. 2018
- [Background] Phadke A, Bedekar N, Shyam A, Sancheti P. Effect of muscle energy technique and static stretching on pain and functional disability in patients with mechanical neck pain: A randomized controlled trial. Hong Kong Physiother J. 2016 Apr 14;35:5-11. doi: 10.1016/j.hkpj.2015.12.002. eCollection 2016 Dec. PMID 30931028
- [Background] Mahajan, R., C. Kataria, and K. Bansal, Comparative effectiveness of muscle energy technique and static stretching for treatment of subacute mechanical neck pain. Int J Health Rehabil Sci, 2012. 1(1): p. 16-21
- [Background] Crothers AL, French SD, Hebert JJ, Walker BF. Spinal manipulative therapy, Graston technique(R) and placebo for non-specific thoracic spine pain: a randomised controlled trial. Chiropr Man Therap. 2016 May 16;24:16. doi: 10.1186/s12998-016-0096-9. eCollection 2016. PMID 27186365
- [Background] • Gupta, S., P. Jaiswal, and D. Chhabra, A comparative study between postisometric relaxation and isometric exercises in non-specific neck pain. Journal of exercise science and physiotherapy, 2008. 4(2): p. 88
- [Background] Joshi R, Rathi M. Effect of Muscle Energy Technique versus Positional Release Technique on Pain and Functions in Patients with Trapezitis-A Comparative Study. Internafional Journal of Science and Research. 2017;6:2113-5.
- [Background] • Kumari C, Sarkar B, Banerjee D, Alam S, Sharma R, Biswas A. Efficacy of muscle energy technique as compared to proprioceptive neuromuscular facilitation technique in chronic mechanical neck pain: A randomized controlled trial. Int J Health Sci Res. 2016; 6:152-61.